CLINICAL TRIAL: NCT06111859
Title: Real-time Elastography for Non-invasive Assessment of Liver Fibrosis and Fat Quantification Techniques for Assessment of Fatty Change in Chronic Liver Disease
Brief Title: Effectiveness of Ultrasound in Liver Stiffness and Fat Quantification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Samsung Medison (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 212836
Record Dates: First submitted 2023-09-14; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Liver Disease Chronic; Fibrosis, Liver; Liver Steatoses; Liver Fat; NAFLD; NASH With Fibrosis; Hepatitis
Keywords: Elastography; Fat Quantification Liver; Chronic liver disease; NAFLD; MAFLD; Hepatitis; Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver; Non-alcoholic Fatty Liver Disease; Hepatitis; Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver Biopsy Cohort (Experimental)
  Interventions: Diagnostic Test: Ultrasound based Elastography and fat quantification

INTERVENTIONS:
Diagnostic Test: Ultrasound based Elastography and fat quantification — Correlation of ultrasound-based elastography and fat quantification on liver biopsy

SUMMARY:
Liver stiffness is a marker for scarring of the liver, which occurs after damage from various liver conditions. Scarring prevents normal liver function and can lead to liver failure. Fatty liver is a common cause of liver damage and can contribute to scarring.

Currently, liver biopsy serves as the 'gold standard' for assessing the degree of liver scarring and fatty infiltration, guiding treatment decisions. However, liver biopsy poses a significant risk of death and unpleasant side effects, including internal bleeding and pain. Moreover, due to the small sample of liver tissue obtained during the biopsy, the results can be misleading and may not provide an accurate overview of the liver's health. Therefore, there is an unmet need for a non-invasive method of measuring liver stiffness and fat content.

Ultrasound-based methods utilize various properties of ultrasound waves to assess liver stiffness and fat levels. This study aims to recruit 100-120 patients with chronic liver disease. The investigators will assess liver stiffness and fat levels during patients' hospital visits for routine scans, biopsies, or clinic appointments. The resulting measurements of liver stiffness and fat obtained through ultrasound-based methods will be compared to patients' routine liver biopsies, routine FibroScan results (another non-invasive method routinely used in clinical care to assess patients' liver stiffness), and other non-invasive severity scores (calculated from results obtained from patients' routine blood tests, providing an overview of the extent of liver damage).

DETAILED DESCRIPTION:
Elastography and fat quantification techniques are imaging methods integrated into the normal B-mode ultrasound. These techniques are extremely safe, with no additional risk compared to a normal ultrasound study. The advantage of using liver elastography/fat techniques to assess the degree of liver fibrosis/fatty change is that the techniques are non-invasive (no needles or biopsies) with higher patient acceptance and compliance. Shear wave elastography is a non-invasive technique that can quantify liver stiffness by measuring the speed of shear waves in the tissue of interest. Early studies have shown that the speed of the shear wave is closely associated with different stages of liver fibrosis. It has also been shown that the measurements can be reproduced by different investigators. Fatty changes, assessed by measurements called TAI, TSI, and EzHRI, are in the early stages of investigation and are proving to be robust. Early studies are mostly performed using elastography have been investigated using Fibroscan (vibration shear wave generator) techniques, and to a lesser extent using point and 2-D shearwave elastography. Fat quantification is also undertaken on the Fibroscan system, producing a Controlled Attenuation Parameter (CAP) measurement which can be correlated both to the fat quantification methods and biopsy result. The investigators have, through a previous project, demonstrated that liver stiffness, using point shear wave, on other machines can accurately identify different stages of liver fibrosis. The investigators would like to extend the study to include a further commercially available machine, namely Samsung RS85 Prestige, to study its diagnostic accuracy of point and 2-D elastography and the fat quantification techniques. As more machines with similar capabilities for stiffness and fat assessment become available, data would be collected from these also. In addition, this study will enrich scientific evidence in terms of how accurate elastography/fat assessment is as a method of measuring liver stiffness/fatty change and hopefully reduce the need to perform liver biopsy in the future.

ELIGIBILITY:
Inclusion Criteria:

1. >=18 years old
2. Male or Female
3. Suspected chronic liver disease based on clinical history, serum biochemistry, prior imaging or prior liver biopsy
4. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Liver transplantation within the last six months
2. Suspected or known acute liver disease
3. Focal liver lesion(s)
4. Age <18 years old
5. Pregnant women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-01-02 (Estimated); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of liver elastography compared to histological staging | 3 years
  Comparison of ultrasound elastography measures and biopsy based fibrosis scores
Diagnostic accuracy of liver fat quantification compared to histological assessment | 3 years
  Comparison of ultrasound fat quantification measures and biopsy based fat percentages

CONTACTS AND LOCATIONS:
Locations (1):
- Nuran Seneviratne, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No